CLINICAL TRIAL: NCT03113604
Title: Analysis of the Role of Hepatocyte SLAMF3 Receptor and Drug Resistance Proteins (MDR) in Resistance to Treatment With Sorafenib in CHC Patients
Acronym: SLAMF3
Status: Withdrawn | Type: Observational
Why Stopped: The study has been stopped because no one is
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2015_843_0021
Record Dates: First submitted 2017-04-10; First posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Hepatocyte Receptor; Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with untreated CHC not sorafenib
  Interventions: Other: Study on samples of tumor and peri-tumor tissues from patients with hepatocellular carcinoma
- Patients with non-sorafenib CHC
  Interventions: Other: Study on samples of tumor and peri-tumor tissues from patients with hepatocellular carcinoma
- Patients with CHCs responding to sorafenib
  Interventions: Other: Study on samples of tumor and peri-tumor tissues from patients with hepatocellular carcinoma

INTERVENTIONS:
Other: Study on samples of tumor and peri-tumor tissues from patients with hepatocellular carcinoma — Retrospective study of samples of tumor and peri-tumor tissues from patients with hepatocellular carcinoma (HCC): three groups of samples will be selected:
  Group 1: Tumor and peri-tumor tissue samples from patients with non-treated sorafenib CHC (surgical resection or other) Group 2: Tumor and peri-tumor tissue samples from tumor and peritumor tissues of patients not responding to sorafenib treatment Group 3: samples from patients responding to treatment with sorafenib

SUMMARY:
Primary liver cancer or hepatocellular carcinoma (HCC) is the 7th most common cancer in humans; 9th in women (figures from the Association for Research against Cancer ARC). This cancer is a major public health problem on a global scale. Patients, whose diagnosis is often late, are at advanced stages of the pathology, even those who benefit from locoregional treatments have a poor prognosis and suffer from a lack of curative therapeutic strategies. CHC is highly refractory to cytotoxic chemotherapy and so far the response rates to conventional systemic chemotherapy has provided a clinical benefit where survival was prolonged by more than 25% in patients with advanced CHC. Further efforts are needed to effectively manage HCC. Knowledge of the mechanisms regulating proliferation and inhibiting the sensitivity of transformed cells to apoptosis is the key to the development of more effective therapeutic strategies.

Several new therapies, called targeted therapies, are tested in clinical trials. Currently, the most effective molecular agent for targeting the Raf pathway is sorafenib capable of also inhibiting tyrosine kinases of VEGFR and PDGFR. Sorafenib, a multikinase inhibitor, decreases the proliferation of tumor cells in vitro that inhibit the activity of targets present in tumor cells (CRAF, BRAF, V600E BRAF, c-KIT, and FLT-3) and tumor vascularization VEGFR-2, VEGFR-3, and PDGFR-beta). Despite the real benefit of this treatment, its efficacy (three months of overall survival) and its indication remain limited to Child-Pugh A, WHO 0-2 patients in whom curative treatment is contraindicated. In addition, several patients have resistance to Sorafenib and thus find themselves in therapeutic failure, thus limiting the therapeutic choice for these patients.

Resistance to treatment with Sorafenib limits the therapeutic choice. The mechanisms responsible for this resistance remain to be elucidated. Drug resistance proteins, MDR Multi-Drug Resistance, is a family of molecules whose expression increases in the cancer cell and ensures the repression of chemotherapy molecules outside the target cancer cell. This family includes the proteins ABCG2, MDR and MRP1. Our in vitro studies show that treatment of CHC Huh-7 cells with Sorafenib (10 mM) induces the specific expression of the transcripts of the MRP-1 protein without any effect on the expression of the ABCG2 and MDR protein. In addition, sorafenib has an effect on the expression of hepatocyte SLAMF3 receptor transcripts, a receptor recently identified in hepatocyte tissue. Indeed, it has been shown that the expression of SLAMF3 is lowered in the cancerous tissue compared to the healthy tissue and that the reintroduction of a strong expression in the cancer cell inhibits its proliferation by inhibiting the MAPK Erk pathway, Cancer cells to apoptosis and inhibits the uptake of tumor masses in the Nude mouse (I. Marcq, et al., 2013).

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age,
* Diagnosis of hepatocellular carcinoma (histological or non-invasive criteria of Barcelona),

Group 1: Tumor and peri-tumor tissue samples from patients with untreated CHCs sorafenib

- Patients who received treatment other than sorafenib (chemo-embolization, radiofrequency, resection, ...),

Group 2: Tumor and peri-tumor tissue samples from patients with non-sorafenib CHC

* Patients treated with sorafenib,
* Patients not responding to treatment with sorafenib

Group 3: Tumor and peri-tumor tissue samples from patients with CHCs responding to sorafenib

* Patients treated with sorafenib,
* Patients responding to treatment with sorafenib

Exclusion Criteria:

* Age <18 years,
* Patients who do not have liver biopsy specimens (PBH) available at the tumor bank,
* Patients who have refused to use their samples for biomedical research,
* Pregnancy and breast feeding

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Group 1: Tumor and peri-tumor tissue samples from patients with non-treated sorafenib CHC (surgical resection or other) Group 2: Tumor and peri-tumor tissue samples from tumor and peritumor tissues of patients not responding to sorafenib treatment Group 3: samples from patients responding to treatment with sorafenib
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-11-20 (Actual); Primary Completion 2016-11-20 (Actual); Study Completion 2016-11-20 (Actual)

PRIMARY OUTCOMES:
Rate of expression of SLAM3 and MDR transcripts, correlation with the responder status or not with Sorafenib | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France